CLINICAL TRIAL: NCT01697449
Title: An Observational Study of Avastin (Bevacizumab) in Patients With Metastatic Colorectal Cancer (RELEVANT)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21889
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective observational study will evaluate the safety and efficacy of Avastin (bevacizumab) in patients with metastatic colorectal cancer. Data will be collected from patients receiving Avastin in combination with chemotherapy according to registered indication in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Metastatic colorectal cancer
* Prescribed to receive Avastin according to registered indication

Exclusion Criteria:

* Patients not eligible for Avastin treatment according to the Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer initiated on Avastin in combination with chemotherapy
Sampling Method: Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2009-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Serbia (4):
  - Belgrade
  - Kamenitz
  - Kragujevac
  - Niš

RESULTS

PARTICIPANT FLOW:
Groups:
- Colorectal Cancer (CRC) Cohort: Participants with metastatic CRC (resectable/unresectable at baseline) received bevacizumab in combination with chemotherapy according to registered indication in routine clinical practice until progression of disease, unacceptable toxicity, lost to follow up, death, or withdrawal of informed consent.
Period: Overall Study
Arm/Group | Colorectal Cancer (CRC) Cohort
Started | 191
Completed | 101
Not Completed | 90
Not completed — Disease progression | 47
Not completed — Adverse Event | 7
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — Death | 2
Not completed — Other | 1
Not completed — Missing | 25

BASELINE CHARACTERISTICS:
Population: Included all participants who were enrolled in the study.
Groups:
- CRC Cohort: Participants with metastatic CRC (resectable/unresectable at baseline) received bevacizumab in combination with chemotherapy according to registered indication in routine clinical practice until progression of disease, unacceptable toxicity, lost to follow up, death, or withdrawal of informed consent.
Arm/Group | CRC Cohort
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.31 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least One Adverse Event (AE)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug.
Time Frame: Up to 65 months
Population: All participants who received at least 1 dose of study drug and underwent subsequent safety assessment were considered for the safety analysis.
Measure: Number; unit: percentage of participants
Arm/Group | CRC Cohort
Number analyzed (Participants) | 191
percentage of participants | 15.2

2. Secondary Outcome: Percentage of Participants With Clinical Benefit of Complete Response [CR], Partial Response [PR] or Stable Disease [SD] Per Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Per RECIST, CR was defined as the disappearance of all target and non-target lesions and normalization of tumor marker level; PR was defined as at least a 30 percentage (%) decrease in the sum of the longest diameter of target lesions, taking as reference the screening sum longest diameter; SD for target lesions was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started and SD for non-target lesions defined as persistence of 1 or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits. PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions (target and nontarget lesions) or the unequivocal progression of existing non-target lesions.
Time Frame: Up to 65 months
Population: All participants who received at least 1 dose of study drug were included in this analysis.
Measure: Number; unit: percentage of participants
Groups:
- Resectable/Potentially Resectable CRC at Baseline: Participants with resectable metastatic CRC at baseline received bevacizumab in combination with chemotherapy according to registered indication in routine clinical practice until progression of disease, unacceptable toxicity, lost to follow up, death, or withdrawal of informed consent..
- Unresectable CRC at Baseline: Participants with unresectable metastatic CRC at baseline received bevacizumab in combination with chemotherapy according to registered indication in routine clinical practice until progression of disease, unacceptable toxicity, lost to follow up, death, or withdrawal of informed consent..
Arm/Group | Resectable/Potentially Resectable CRC at Baseline | Unresectable CRC at Baseline
Number analyzed (Participants) | 162 | 29
percentage of participants | 72 | 69

3. Secondary Outcome: Percentage of Participants Who Were Resectable Postbaseline Among the Participants Who Were Unresectable at Baseline
Time Frame: Up to 65 months
Population: Included participants whose CRC was identified as unresectable at baseline.
Measure: Number; unit: percentage of participants
Groups:
- Unresectable: Participants with unresectable metastatic CRC at baseline received bevacizumab in combination with chemotherapy according to registered indication in routine clinical practice until progression of disease, unacceptable toxicity, lost to follow up, death, or withdrawal of informed consent..
Arm/Group | Unresectable
Number analyzed (Participants) | 29
percentage of participants | 34.5

4. Secondary Outcome: Percentage of Participants With Disease Progression or Death
Description: Per RECIST, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions (target and nontarget lesions) or the unequivocal progression of existing non-target lesions.
Time Frame: Up to 65 months
Population: Included participants who received at least 1 dose of study drug and had postbaseline tumor assessment.
Measure: Number; unit: percentage of participants
Arm/Group | CRC Cohort
Number analyzed (Participants) | 170
percentage of participants | 76.5

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of informed consent until the date when the participant had progression of disease or died due to any cause. Participants who left the study for reasons other than progression of the disease were censored at the time of their last tumor assessment. Per RECIST, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions (target and non-target lesions) or the unequivocal progression of existing non-target lesions.
Time Frame: Up to 65 months
Population: Included participants who received at least 1 dose of study drug and had postbaseline tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CRC Cohort
Number analyzed (Participants) | 170
months | 9 [8.24 to 9.75]

ADVERSE EVENTS:
Time Frame: Up to 65 months
Arm/Group | CRC Cohort
Serious Adverse Events (participants affected / at risk) | 23/191
Other Adverse Events (participants affected / at risk) | 9/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CRC Cohort (N=191)
Tuberculosis (Infections and infestations) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Peripheral Artery Thrombosis (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Fatigue (General disorders) | 2
Impaired Healing (General disorders) | 1
Sudden Death (General disorders) | 1
Body Temperature Increased (Investigations) | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CRC Cohort (N=191)
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypertension (Vascular disorders) | 1
Disease progression (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Proteinuria (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.